CLINICAL TRIAL: NCT05337579
Title: Combined Effects of Exercise Breaks and Rest Breaks on Fatigue and Musculoskeletal Discomfort in Static Workstation Office Workers
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Foundation University Islamabad (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: FUI/CTR/2022/6
Record Dates: First submitted 2022-04-14; First posted 2022-04-20 (Actual); Last update posted 2022-04-20 (Actual); Status verified 2022-04

CONDITIONS: Musculoskeletal Pain
MeSH Terms: conditions — Musculoskeletal Pain

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Supplemental Rest Breaks (Active Comparator)
  Interventions: Other: Supplemental Micro Breaks
- Exercise Breaks (Active Comparator)
  Interventions: Procedure: Exercise Breaks
- Supplemental Rest and Exercise Breaks (Experimental)
  Interventions: Other: Supplemental Micro Breaks; Procedure: Exercise Breaks

INTERVENTIONS:
Other: Supplemental Micro Breaks — Supplemental Micro Breaks, of 30 seconds after every 15 minutes of working on a static computer workstation in addition to the two 'Conventional Rest Breaks' of 15 minutes twice a day during the work hours
  Arms: Supplemental Rest Breaks; Supplemental Rest and Exercise Breaks
Procedure: Exercise Breaks — Exercise Breaks, of 10 minutes, twice a day during the work hours, in addition to the two 'Conventional Rest Breaks' of 15 minutes, twice a day during the work hours.
  Arms: Exercise Breaks; Supplemental Rest and Exercise Breaks

SUMMARY:
Musculoskeletal discomfort and work fatigue has enormous impact on quality of personal and professional life and increases health related economic burden on country due to increased cost of healthcare and reduced productivity in work. Upper limb and neck pain complains are the most frequent when evaluated in computer workers. The incidence of musculoskeletal discomfort in office workers is as high as 50%. While fatigue is also common due to its high prevalence and its relationship with dysfunctional disorders in office workers. The objective of this study is to compare and determine the effects of exercise breaks, rest breaks and exercise along with rest breaks on Fatigue and Musculoskeletal discomfort in static workstation office workers

ELIGIBILITY:
Inclusion Criteria:

* Both male and female
* Age: 25-45 years
* Those static workstation office workers using computer for at least 6 hours per day.
* Static workstation office workers screened by ROSA.

Exclusion Criteria:

* Discomfort from non-musculoskeletal origin
* Recent history of trauma and receiving any kind of treatment for the current condition.
* Severe orthopedic disease
* Any mental and physiological illness that could interfere in the exercise.

Ages: 25 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Estimated)
Dates: Start 2022-04-22 (Estimated); Primary Completion 2022-08-22 (Estimated); Study Completion 2022-08-30 (Estimated)

PRIMARY OUTCOMES:
Musculoskeletal Discomfort | 5th week
  Cornell Musculoskeletal Discomfort questionnaire will be used to measure discomfort. A higher score means greater discomfort.
Fatigue | 5th week
  Chalder fatigue scale will be used to measure fatigue. A higher score means greater discomfort.

CONTACTS AND LOCATIONS:
Locations (1):
- Foundation University, Islamabad, Pakistan

IPD SHARING:
Plan to Share IPD: No